CLINICAL TRIAL: NCT04232189
Title: Serum Concentrations of Pregnancy-associated Proteins for Assessment of Gestational Age Before Abortion
Status: Terminated | Type: Observational
Why Stopped: COVID 19 related recruitment problems
Sponsor: Gynuity Health Projects (Other)
Collaborators: Family Planning Associates Medical Group, LTD (Other); Planned Parenthood of Greater New York (Other); Presidential Women's Center (Unknown)
Responsible Party: Sponsor
Other Study IDs: 8003
Record Dates: First submitted 2020-01-14; First posted 2020-01-18 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: Pregnancy
Keywords: placental protein; gestational age; abortion

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Serum and urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — no intervention, just specimen collection

SUMMARY:
This will be a case-series multicenter study enrolling 800 pregnant people. Serum will be collected from people seeking abortion and assayed at a qualified laboratory.

DETAILED DESCRIPTION:
Knowledge of gestational age (GA) is essential for guiding abortion care. In 2016, Gynuity Health Projects (GHP) launched a portfolio of research that aims to explore the possibility of developing a blood or urine test for this purpose.The goal of the present study is to validate initial study findings (protocol 8000) in a larger population of people seeking abortion.

Staff will obtain a serum specimen from each participant before any cervical manipulation is performed and before any abortifacient drug is administered. The site will send the specimens to a central facility for storage until assay. Serum assays for PAPP-A and possibly other proteins will be performed at a selected laboratory by qualified experts.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant and seeking medical or surgical abortion
* Has had or will have an ultrasound on the day of study enrollment or earlier during the current pregnancy
* Able to provide blood and urine specimens before any trans-cervical procedure or mifepristone ingestion
* Not previously enrolled in this study

Exclusion Criteria:

* Does not meet Inclusion Criteria

Sex: Female
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant people seeking abortion at multiple clinics that provide abortion through at least 18 weeks of gestation.
Sampling Method: Non-Probability Sample
Enrollment: 275 (Actual)
Dates: Start 2019-11-12 (Actual); Primary Completion 2020-04-14 (Actual); Study Completion 2020-04-14 (Actual)

PRIMARY OUTCOMES:
Negative Predictive Value 70 days | 1 day
  Negative Predictive Value of Prespecified Protein Concentration in Serum for Predicting a GA of ≤70 days is >95%
Negative Predictive Value 105 days | 1 day
  Negative Predictive Value of Prespecified Protein Concentration in Serum for Predicting a GA of ≤105 days is >95%

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth G Raymond, MD, Principal Investigator — Gynuity Health Projects
Locations (3):
- United States (3):
  - Presidential Women's Center, West Palm Beach, Florida
  - Family Planning Associates, Chicago, Illinois
  - Planned Parenthood of New York City, New York, New York

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Frye LJ, Buhimschi IA, Raymond EG, Zhao G, Winikoff B. PAPP-A as a screening tool for assessment of gestational age before medication abortion in an intended-use population. Biomark Med. 2023 Jan;17(2):73-85. doi: 10.2217/bmm-2022-0653. Epub 2023 Apr 11. PMID 37038980